CLINICAL TRIAL: NCT00549146
Title: Multi-centre, DB, R and Stratified Parallel Group Study to Compare the Efficacy and Safety of FP 500mcg Bid vs. SRT 50/250mcg Via Diskus in COPD Pts With Partial Reversible Obstruction
Brief Title: Treatment Of Partial Reversible Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCO40055
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: reversibility; COPD; lung function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol 250/50 DISKUS combination product
Drug: fluticasone propionate DISKUS 500mcg
  Other Names: fluticasone propionate/salmeterol 250/50 DISKUS combination product

SUMMARY:
Relatively little information is available about the effects of salmeterol/fluticasone combination and fluticasone alone in COPD patients with a partial reversible pulmonary obstruction. The purpose of this study is to compare the effects of salmeterol/fluticasone combination with fluticasone alone delivered via Diskus/ACCUHALER inhaler in subjects with COPD on lung function over a 1 year period.

DETAILED DESCRIPTION:
Multi-centre, double-blind, randomised and stratified parallel group study to compare the efficacy and safety of fluticasone propionate 500 mcg bd versus salmeterol/fluticasone combination 50/250 mcg bd both via Diskus inhaler during 1 year in Chronic Obstructive Pulmonary Disease(COPD) patients with a partially reversible obstruction.

ELIGIBILITY:
Inclusion criteria:

* Established history of chronic obstructive pulmonary disease (COPD).
* Lung function parameters: FEV1/FVC ratio < 70%, FEV1 between 80% and 30% predicted, a reversibility of airway obstruction of 12% of the initial value with a minimum of 200 mL.
* Signed and dated informed consent.

Exclusion criteria:

* History of asthma or allergy.
* Unstable COPD in the 3 months before the study.
* Interference of non-pulmonary medication or diseases with COPD outcome parameters.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2003-11 (Actual); Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Difference in efficacy of a 12 months treatment with salmeterol/fluticasone combination versus fluticasone on lung function (FEV1) as percentage predicted.

SECONDARY OUTCOMES:
Reversibility of lung function with salbutamol and on Forced Vital capacity (FVC), TLC, FRC, FVC, Inspiration capacity(IC), Forced Inspiratory Volume in 1 second (FIV1) and Maximum mid-Expiratory Flow (MEF50).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- Netherlands (15):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Drachten
  - GSK Investigational Site, Haarlem
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Hengelo
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Leeuwarden
  - GSK Investigational Site, Meppel
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Sneek
  - GSK Investigational Site, Utrecht
  - GSK Investigational Site, Voerendaal